CLINICAL TRIAL: NCT02333799
Title: A Phase 3 Open-label Trial Assessing the Safety and Efficacy of Bedaquiline Plus PA-824 Plus Linezolid in Participants With Pulmonary Infection of Either XDR-TB or Treatment Intolerant / Non-responsive MDR-TB.
Brief Title: A Phase 3 Trial Assessing Safety and Efficacy of B-Pa-L in Participants With DR-TB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nix-TB-(B-L-Pa)
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; MDR-TB; XDR-TB; Multi-drug resistant; Extensively drug resistant; Bedaquiline; PA-824; Linezolid; TB; Pretomanid; TMC-207; NiX-TB
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis; Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis | interventions — bedaquiline; pretomanid; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bedaquiline + PA-824 + Linezolid (Experimental): bedaquiline 400 mg once daily for 2 weeks then 200mg 3 times per week plus PA-824 200mg once daily plus linezolid 1200mg once daily.
  A reduction in the dose of linezolid (to either 600 mg qd or 300 mg qd), or temporary cessation of linezolid (due to a linezolid-specific toxicity), or of the full regimen per Investigator discretion was allowed for suspected drug related toxicity. Re-introduction of the regimen could be considered post a cessation not greater than 35 consecutive days.
  If participants had toxicity events related to linezolid prohibiting further treatment with that drug, they could remain on the bedaquiline and pretomanid study IMP if they received the initial total of 1200 mg daily dose of linezolid for at least the first 4 consecutive weeks of treatment and they were smear negative, or with trace/scanty results and judged to be clinically improving by the Investigator.
  Interventions: Drug: Bedaquiline; Drug: PA-824; Drug: Linezolid

INTERVENTIONS:
Drug: Bedaquiline — 100mg tablets
  Other Names: B; TMC-207
Drug: PA-824 — 200mg tablets
  Other Names: Pa; pretomanid
Drug: Linezolid — Scored 600mg tablets
  Other Names: L; Lin

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability and pharmacokinetics of bedaquiline plus PA-824 plus linezolid after 6 months of treatment (option for 9 months for participants who remain culture positive at month 4) in participants with either pulmonary extensively drug resistant tuberculosis (XDR-TB), treatment intolerant or non-responsive multi-drug resistant tuberculosis (MDR-TB).

DETAILED DESCRIPTION:
Up to 200 male and female participants aged 14 and over with confirmed sputum positive for M.tb. in culture pulmonary XDR-TB, or with pulmonary MDR-TB with a documented intolerability or non-response to the best treatment available for 6 months or more will be enrolled.

All participants will have up to a maximum of 9 days for screening, receive 6 months of treatment, and have followup visits performed 1 and 2 months after treatment completion and every 3 months after study treatment completion for 24 months. If a participant is culture positive or revert to being culture positive between Month 4 and Month 6 visits and their clinical condition suggests they may have ongoing TB infection, they may have treatment extended to 9 months (with 24 months of Follow Up) or be withdrawn from the study.

Participants who withdraw after <14 days of IMP should attend an Early Withdrawal visit. Participants who withdraw after >15 days of IMP should return for an Early Withdrawal visit and follow-up visits at 3, 6 and 24 months after their last dose of IMP to check for survival, SAEs and resolution of TB symptoms.

ELIGIBILITY:
Key Inclusion Criteria

1. Provide written, informed consent prior to all trial-related procedures (if under 18, include consent of legal guardian).
2. Body weight of ≥35 kg (in light clothing and no shoes).
3. Male or female, aged 14 years or above.
4. Subjects with one of the following pulmonary TB conditions (WHO definitions prior to 2021):

   a. Extensively Drug Resistant Tuberculosis (XDR-TB) with

   i. documented culture positive (for M.tb.) results within 3 months prior to screening or M.tb. confirmed in sputum based on molecular test within 3 months prior to or at screening;

   ii. documented resistance to isoniazid, rifamycins, a fluoroquinolone and an injectable historically at any time or at screening;

   b. Multi-Drug Resistant Tuberculosis (MDR-TB) documented by culture positive results (for M.tb.) within 3 months prior to or at screening with documented non-response to treatment with the best available regimen for 6 months or more prior to enrolment who in the opinion of the Investigator have been adherent to treatment and will be adherent to study regimen;

   c. MDR-TB documented by culture positive (for M.tb.) results within 3 months prior to or at screening who are unable to continue second line drug regimen due to a documented intolerance to:

   i. PAS, ethionamide, aminoglycosides or fluoroquinolones;

   ii. Current treatment not listed above that renders subject eligible for the study in the Investigator's opinion.

6. Chest X-Ray picture (taken within a year prior to screening) consistent with pulmonary TB in the opinion of the Investigator.

Key Exclusion Criteria

1. Karnofsky score < 50 within 30 days prior to entry.
2. Body Mass index (BMI) < 17 kg/m²
3. History of allergy or known hypersensitivity to any of the trial Investigational Medicinal Products or related substances.
4. HIV infected Subjects having a CD4+ count ≤ 50 cells/μL
5. Having participated in other clinical studies with dosing of investigational agents within 8 weeks prior to trial start or currently enrolled in an investigational study that includes treatment with medicinal agents. Subjects who are participating in observational studies or who are in a follow up period of a trial that included drug therapy may be considered for inclusion.
6. Significant cardiac arrhythmia requiring medication.
7. Subjects with the following at Screening:

   1. QTcF interval on ECG >500 msec.
   2. History of additional risk factors for Torsade de Pointes, (e.g., heart failure, hypokalemia, family history of Long QT Syndrome);
   3. Clinically significant ventricular arrhythmias;
   4. Subjects with other cardiac abnormalities that may place them at risk of arrhythmias must be discussed with the sponsor medical monitor before enrolment. Such abnormalities include: Evidence of ventricular pre-excitation (e.g., Wolff Parkinson White syndrome); Electrocardiographic evidence of complete or clinically significant incomplete left bundle branch block or right bundle branch block; Evidence of second or third degree heart block; Intraventricular conduction delay with QRS duration more than 120 msec.
8. Females who have a positive pregnancy test at Screening or already known to be pregnant, breastfeeding, or planning to conceive a child during the study or within 6 months of cessation of treatment. Males planning to conceive a child during the study or within 6 months of cessation of treatment.
9. A peripheral neuropathy of Grade 3 or 4, according to DMID (Appendix 2). Or, subjects with a Grade 1 or 2 neuropathy which is likely to progress/worsen over the course of the study, in the opinion of the Investigator.
10. Concomitant use of Monoamine Oxidase Inhibitors (MAOIs) or prior use within 2 weeks of treatment assignment.
11. Subjects with the following toxicities at Screening as defined by the enhanced Division of Microbiology and Infectious Disease (DMID) adult toxicity table (November 2007):

    a. serum potassium less than the lower limit of normal for the laboratory; b. Hemoglobin level grade 2 or greater (< 8.0 g/dL); c. Platelets grade 2 or greater(<75,000/mm3); d. Absolute neutrophil count (ANC) < 1000/ mm3; e. Aspartate aminotransferase (AST) > 3 x ULN g. Total bilirubin > or = to 2xULN h. Direct bilirubin > ULN i. Serum creatinine level greater than 2 times upper limit of normal j. Albumin <32 g/L

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-03; Primary Completion 2019-01-14 (Actual); Study Completion 2020-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morounfolu Olugbosi, MD, Principal Investigator — Global Alliance for TB Drug Development; Francesca Conradie, MD, Principal Investigator — CHRU Themba Lethu Clinic - Helen Joseph Hospital
Locations (3):
- South Africa (3):
  - Task Applied Science - Brooklyn Chest Hospital, Ysterplaat, Cape Town
  - King DinuZulu Hospital Complex, Sydenham, Durban
  - Sizwe Tropical Disease Hospital, Sandringham, Johannesburg

REFERENCES:
- [Derived] Solans BP, Imperial MZ, Olugbosi M, Savic RM. Analysis of Dynamic Efficacy Endpoints of the Nix-TB Trial. Clin Infect Dis. 2023 Jun 8;76(11):1903-1910. doi: 10.1093/cid/ciad051. PMID 36804834
- [Derived] Imperial MZ, Nedelman JR, Conradie F, Savic RM. Proposed Linezolid Dosing Strategies to Minimize Adverse Events for Treatment of Extensively Drug-Resistant Tuberculosis. Clin Infect Dis. 2022 May 30;74(10):1736-1747. doi: 10.1093/cid/ciab699. PMID 34604901
- [Derived] Conradie F, Diacon AH, Ngubane N, Howell P, Everitt D, Crook AM, Mendel CM, Egizi E, Moreira J, Timm J, McHugh TD, Wills GH, Bateson A, Hunt R, Van Niekerk C, Li M, Olugbosi M, Spigelman M; Nix-TB Trial Team. Treatment of Highly Drug-Resistant Pulmonary Tuberculosis. N Engl J Med. 2020 Mar 5;382(10):893-902. doi: 10.1056/NEJMoa1901814. PMID 32130813
- See also: TB Alliance Website — http://www.tballiance.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening Phase: 143 participants were screened to determine eligibility to participate in the study using inclusion and exclusion criteria within 9 days of scheduled day 1 treatment dosing. 34 participants did not meet treatment criteria and were excluded from further study participation. 109 participants were enrolled in the study and began the treatment phase of the study.
Groups:
- Bedaquiline + PA-824 + Linezolid: Bedaquiline (Days 1 to 14): 400 mg once daily (4 x bedaquiline 100mg tablets); Bedaquiline (Weeks 3 to 26 or 39*): 200 mg three days a week (2 x bedaquiline 100 mg tablets); plus Pretomanid: (Day 1 through weeks 26 or 39*) 200 mg once daily (1 x pretomanid 200 mg tablet); plus Linezolid: (Day 1 through weeks 26 or 39*) 1200 mg daily (1 x linezolid 600 mg tablet twice daily, later amended to 2 x linezolid 600 mg tablets once daily)
  *Note - participants received a minimum of 6 months (week 26) of trial treatment. If participants were culture positive or reverted to being culture positive between month 4 and month 6, and their clinical condition suggested they may have ongoing TB infection, the trial treatment could have been extended to 9 months (week 39).
Period: Treatment Period
Arm/Group | Bedaquiline + PA-824 + Linezolid
Started (All participants were to receive 6 months of treatment, from Day 1 to week 26 (6 months) or Day 1 to week 39 (9 months). Participants that were culture negative moved to the Follow Up Period. If participants were culture positive or reverted to being culture positive between the Month 4 and Month 6 visits, and their clinical condition suggested they may have ongoing TB infection, their Treatment Period could have been extended to 9 months.) | 109
Completed | 102
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Death | 6
Period: 6 Month Follow Up Period
Arm/Group | Bedaquiline + PA-824 + Linezolid
Started | 102
Completed | 100
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Death | 1
Period: 7 to 24 Month Follow Up Period
Arm/Group | Bedaquiline + PA-824 + Linezolid
Started | 100
Completed | 98
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Bedaquiline + PA-824 + Linezolid: bedaquiline 400 mg once daily for 2 weeks then 200mg 3 times per week plus PA-824 200mg once daily plus linezolid 1200mg once daily .
  Bedaquiline: 100mg tablets
  PA-824: 200mg tablets
  Linezolid: Scored 600mg tablets
Arm/Group | Bedaquiline + PA-824 + Linezolid
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 83
  White | 1
  More than one race | 25
  Unknown or Not Reported | 0
Height (cm) [Mean (Standard Deviation); unit: cm] — Population: total number with height recorded
  cm
    number analyzed (Participants) | 108
    (all) | 165.78 (10.408)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 56.95 (15.034)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 20.60 (5.046)
CD4 Count (cells/uL) [Mean (Standard Deviation); unit: cells/uL] — Population: CD4 count for HIV positive patient (with a CD4 count available)
  cells/uL
    number analyzed (Participants) | 51
    (all) | 394.0 (212.00)
Karnofsky Score (%) [Count of Participants; unit: Participants] — Measure Description: Trained clinicians interview participants and grade their ability to perform daily activities using a percent scale where higher scores indicate that the participant is better able to function than lower scores. 100% indicates normal activity with no evidence of disease whereas a score of 70% or lower would indicate that the participant is unable to work and 40% or lower is unable to care for themselves. http://www.npcrc.org/files/news/karnofsky_performance_scale.pdf
  Participants
    100 (Normal, no complaints) | 9
    90 | 50
    80 | 29
    70 | 19
    60 | 2
    50 | 0
    40 | 0
    30 | 0
    20 | 0
    10 | 0
    0 (Dead) | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Treatment Failure (Unfavorable Outcome), Defined as Bacteriologic Failure or Relapse or Clinical Failure (Derived) Through Follow-up Until 6 Months After the End of Treatment.
Description: Bacteriologic failure: During the treatment period, failure to attain culture conversion to negative.
  Bacteriologic relapse: During the follow-up period, failure to maintain culture conversion to negative status in culture, with culture conversion to positive status with a Mycobacterium tuberculosis (M.tb.) strain that is genetically identical to the infecting strain at baseline.
  Clinical failure: A change from protocol-specified tuberculosis (TB) treatment due to treatment failure, retreatment for TB during follow up, or TB-related death.
  Note:
  Culture conversion requires at least 2 consecutive culture negative/positive samples at least 7 days apart.
  Participants who are documented at a visit as unable to produce sputum and who are clinically considered to be responding well to treatment will be considered to be culture negative at that visit.
Time Frame: 6 Months post End of Treatment
Population: Participants deemed unassessable were excluded from the Modified Intent to Treat (MITT) population as per the analysis plan.
Measure: Count of Participants; unit: Participants
Groups:
- Total: Total Participants
- XDR-TB: Extensively Drug-Resistant Tuberculosis (XDR-TB) Population
- TI/NR MDR-TB: Treatment-Intolerant/Nonresponsive Multidrug-Resistant Tuberculosis (TB) Population
Arm/Group | Total | XDR-TB | TI/NR MDR-TB
Number analyzed (Participants) | 107 | 70 | 37
Participants
  Favourable (treatment success) | 98 | 63 | 35
  Unfavourable (treatment failure) | 9 | 7 | 2

2. Secondary Outcome: Proportion of Treatment Failure (Unfavorable Outcome), Defined as Bacteriologic Failure or Relapse or Clinical Failure (Derived) Through Follow-up Until 24 Months After the End of Treatment.
Description: Bacteriologic failure: During the treatment period, failure to attain culture conversion to negative.
  Bacteriologic relapse: During the follow-up period, failure to maintain culture conversion to negative status in culture, with culture conversion to positive status with a Mycobacterium tuberculosis (M.tb.) strain that is genetically identical to the infecting strain at baseline.
  Clinical failure: A change from protocol-specified TB treatment due to treatment failure, retreatment for TB during follow up, or TB-related death.
  Note:
  Culture conversion requires at least 2 consecutive culture negative/positive samples at least 7 days apart.
  Participants who are documented at a visit as unable to produce sputum and who are clinically considered to be responding well to treatment will be considered to be culture negative at that visit.
Time Frame: 24 Months post End of Treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Total: Total Population
- XDR-TB: Extensively Drug-Resistant TB Population
- TI/NR MDR-TB: Treatment-Intolerant/Nonresponsive Multidrug Resistant TB Population
Arm/Group | Total | XDR-TB | TI/NR MDR-TB
Number analyzed (Participants) | 106 | 69 | 37
Participants
  Favourable (treatment success) | 96 | 61 | 35
  Unfavourable (treatment failure) | 10 | 8 | 2

3. Secondary Outcome: Time to Sputum Culture Conversion to Negative Status Through the Treatment Period
Description: Median time (in weeks) to culture negative status (first of 2 negative cultures without an intervening positive culture), MITT analysis.
Time Frame: Day 1 through End of Treatment, approximately 6 to 9 months of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Total | XDR-TB | TI/NR MDR-TB
Number analyzed (Participants) | 88 | 59 | 29
Weeks | 6 [4.1 to 8.1] | 6 [4.1 to 8.3] | 6 [4.0 to 8.1]

4. Secondary Outcome: Proportion of Participants With Sputum Culture Conversion to Negative Status
Description: Proportion of participants with sputum culture conversion to negative status for those positive at baseline at 4, 6, 8, 12, 16, and End of Treatment (26 or 39 weeks)
Time Frame: Week 4, 6, 8, 12, 16, 26, 39
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total | XDR-TB | TI/NR MDR-TB
Number analyzed (Participants) | 90 | 60 | 30
Participants
  Week 4: Negative | 37 | 25 | 12
  Week 4: Positive | 53 | 35 | 18
  Week 4: Died | 0 | 0 | 0
  Week 6: Negative | 57 | 37 | 20
  Week 6: Positive | 32 | 22 | 10
  Week 6: Died | 1 | 1 | 0
  Week 8: Negative | 71 | 46 | 25
  Week 8: Positive | 15 | 10 | 5
  Week 8: Died | 4 | 4 | 0
  Week 12: Negative | 82 | 53 | 29
  Week 12: Positive | 3 | 2 | 1
  Week 12: Died | 5 | 5 | 0
  Week 16: Negative | 83 | 55 | 28
  Week 16: Positive | 1 | 0 | 1
  Week 16: Died | 6 | 5 | 1
  End of Treatment: Negative | 84 | 55 | 29
  End of Treatment: Positive | 0 | 0 | 0
  End of Treatment: Died | 6 | 5 | 1

5. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAEs): adverse events which started or worsened on or after the first trial drug administration up to and including 14 days after the last trial drug administration. Grade I, II, III, IV TEAEs: DMID grade is indicated as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (potentially life-threatening). TEAEs of special interest based on Section 7.3 of the protocol. Liver-related adverse events: any adverse event with a High Level Group Term of HEPATIC AND BILIARY NEOPLASMS BENIGN, HEPATIC AND HEPATOBILIARY DISORDERS, HEPATOBILIARY DISORDERS CONGENITAL, HEPATOBILIARY NEOPLASMS MALIGNANT AND UNSPECIFIED, HEPATOBILIARY INVESTIGATIONS or HEPATOBILIARY THERAPEUTIC PROCEDURES.
Time Frame: Day 1 to 14 days post-End of Treatment
Population: Population analyzed contains all participants who received at least 1 dose of study treatment
Measure: Number; unit: events
Groups:
- HIV - Negative: HIV Status Negative Population
- HIV - Positive: HIV Status Positive Population
- 600 mg BID Linezolid: Bedaquiline (Days 1 to 14): 400 mg once daily (4 x bedaquiline 100mg tablets); Bedaquiline (Weeks 3 to 26 or 39*): 200 mg three days a week (2 x bedaquiline 100 mg tablets); plus Pretomanid: (Day 1 through weeks 26 or 39*) 200 mg once daily (1 x pretomanid 200 mg tablet); plus Linezolid: (Day 1 through weeks 26 or 39*) 1200 mg daily (1 x linezolid 600 mg tablet twice daily)
- 1200 mg QD Linezolid: Bedaquiline (Days 1 to 14): 400 mg once daily (4 x bedaquiline 100mg tablets); Bedaquiline (Weeks 3 to 26 or 39*): 200 mg three days a week (2 x bedaquiline 100 mg tablets); plus Pretomanid: (Day 1 through weeks 26 or 39*) 200 mg once daily (1 x pretomanid 200 mg tablet); plus Linezolid: (Day 1 through weeks 26 or 39*) 1200 mg daily (2 x linezolid 600 mg tablets once daily)
- Total: Total Trial Population
  Bedaquiline (Days 1 to 14): 400 mg once daily (4 x bedaquiline 100mg tablets); Bedaquiline (Weeks 3 to 26 or 39*): 200 mg three days a week (2 x bedaquiline 100 mg tablets); plus Pretomanid: (Day 1 through weeks 26 or 39*) 200 mg once daily (1 x pretomanid 200 mg tablet); plus Linezolid: (Day 1 through weeks 26 or 39*) 1200 mg daily (1 x linezolid 600 mg tablet twice daily, later amended to 2 x linezolid 600 mg tablets once daily)
  *Note - participants received a minimum of 6 months (week 26) of trial treatment. If participants were culture positive or reverted to being culture positive between month 4 and month 6, and their clinical condition suggested they may have ongoing TB infection, the trial treatment could have been extended to 9 months (week 39).
Arm/Group | HIV - Negative | HIV - Positive | 600 mg BID Linezolid | 1200 mg QD Linezolid | Total
Number analyzed (Participants) | 53 | 56 | 44 | 65 | 109
events
  Any TEAE | 658 | 633 | 491 | 800 | 1291
  TEAE Leading To Death | 5 | 5 | 6 | 4 | 10
  Serious TEAE (Including Death) | 16 | 20 | 24 | 12 | 36
  TEAE Leading To Early Trial Withdrawal | 5 | 6 | 7 | 4 | 11
  TEAE Leading To Discontinuation Of One Or All Drugs in the Trial Regimen (Per Investigator) | 16 | 23 | 19 | 20 | 39
  TEAE Leading To Interruption Of Trial Drug | 40 | 41 | 46 | 35 | 81
  Grade III and/or IV TEAE | 49 | 77 | 65 | 61 | 126
  Drug-Related TEAE | 387 | 319 | 298 | 408 | 706
  Serious Drug-Related TEAE | 5 | 7 | 9 | 3 | 12
  TEAE of Special Interest | 157 | 158 | 132 | 183 | 315
  Liver-Related TEAE | 27 | 38 | 27 | 38 | 65
  Drug-Related and Liver-Related TEAE | 22 | 33 | 23 | 32 | 55
  Serious Liver-Related TEAE | 1 | 0 | 0 | 1 | 1

6. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs) of Special Interest
Description: Treatment-emergent adverse events (TEAEs): Defined as adverse events which started or worsened on or after the first trial drug administration up to and including 14 days after the last trial drug administration. TEAEs of special interest: Identified by prespecified SMQ codes as confirmed by TB Alliance.
  Section 7.3 of the protocol specified the "Monitoring and Safety for Specific Toxicities" and are presented here as TEAEs of special interest. These specific toxicities of interest were based on nonclinical toxicology findings of concern for any of the 3 trial drugs, or from identified toxicities based on the IBs for pretomanid and bedaquiline, on the product label for linezolid and literature reports of linezolid long-term toxicity.
Time Frame: Day 1 to 14 days post-End of Treatment
Population: The Safety analysis population is defined as all participants who received at least 1 administration of trial treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Bedaquiline + PA-824 + 600 mg BID Linezolid: Population of Bedaquiline + PA-824 + 600 mg BID Linezolid
- Bedaquiline + PA-824 + 1200 mg QD Linezolid: Population of Bedaquiline + PA-824 + 1200 mg QD Linezolid
Arm/Group | HIV - Negative | HIV - Positive | Bedaquiline + PA-824 + 600 mg BID Linezolid | Bedaquiline + PA-824 + 1200 mg QD Linezolid | Total
Number analyzed (Participants) | 53 | 56 | 44 | 65 | 109
Participants
  Peripheral Neurpoathy | 44 | 44 | 33 | 55 | 88
  Haematopoietic Cytopenias | 22 | 30 | 25 | 27 | 52
  Haematopoietic Erythropenia | 16 | 24 | 20 | 20 | 40
  Haematopoietic Leukopenia | 2 | 10 | 5 | 7 | 12
  Haematopoietic Thrombocytopenia | 3 | 3 | 4 | 2 | 6
  Haematopoietic Cytopenias Affecting More Than One Type of Blood Cell | 4 | 1 | 4 | 1 | 5
  Hepatic Disorders | 16 | 26 | 19 | 23 | 42
  Drug-Related Hepatic Disorders - Comprehensive Search | 16 | 26 | 19 | 23 | 42
  Liver-Related Investigations, Signs, and Symptoms | 15 | 25 | 17 | 23 | 40
  Cholestasis and Jaundice of Hepatic Origin | 2 | 3 | 4 | 1 | 5
  Drug-Related Hepatic Disorders - Severe Events Only | 1 | 1 | 2 | 0 | 2
  Hepatic Failure, Fibrosis and Cirrhosis and Other Liver Damage-Related Conditions | 1 | 1 | 2 | 0 | 2
  Optic Nerve Disorders | 9 | 5 | 4 | 10 | 14
  Cardiac Arrhythmias | 5 | 7 | 2 | 10 | 12
  Cardiac Arrhythmia Terms (Incl. Bradyarrhythmias and Tachyarrhythmias) | 3 | 4 | 0 | 7 | 7
  Bradyarrhythmias (Incl. Conduction Defects and Disorders of Sinus Node Function) | 2 | 4 | 0 | 6 | 6
  Conduction Defects | 2 | 4 | 0 | 6 | 6
  Disorders of Sinus Node Function | 1 | 0 | 0 | 1 | 1
  Tachyarrhythmias (Incl. Supraventricular and Ventricular Tachyarrhythmias) | 1 | 0 | 0 | 1 | 1
  Supraventricular Tachyarrhythmias | 1 | 0 | 0 | 1 | 1
  Arrhythmia-Related Investigations, Signs, and Symptoms | 3 | 3 | 2 | 4 | 6
  Rhabdomyolysis/Myopathy | 8 | 3 | 3 | 8 | 11
  Lactic Acidosis | 5 | 3 | 2 | 6 | 8
  Acute Pancreatitis | 1 | 2 | 3 | 0 | 3
  Convulsions | 1 | 1 | 2 | 0 | 2

7. Secondary Outcome: Incidence of Nervous System Disorders - Peripheral Neuropathy Events Grouped
Description: Treatment-emergent adverse events (TEAEs): Defined as adverse events which started or worsened on or after the first trial drug administration up to and including 14 days after the last trial drug administration.
  #: Indicates TEAEs of special interest. TEAEs of special interest: Identified by pre-specified SMQ codes as confirmed by TB Alliance. Adverse events in System Organ Class "NERVOUS SYSTEM DISORDERS" are presented into the table. Preferred term "PERIPHERAL NEUROPATHY" was a grouping of terms "PERIPHERAL SENSORY NEUROPATHY", "NEUROPATHY PERIPHERAL", "PARAESTHESIA", "HYPOAESTHESIA", "PERIPHERAL MOTOR NEUROPATHY", "BURNING SENSATION", "HYPOREFLEXIA" and "PERIPHERAL SENSORIMOTOR NEUROPATHY".
Time Frame: Day 1 to 14 days post-End of Treatment
Population: The Safety analysis population is defined as all participants who received at least 1 administration of trial treatment.
Measure: Number; unit: events
Arm/Group | HIV - Negative | HIV - Positive | Bedaquiline + PA-824 + 600 mg BID Linezolid | Bedaquiline + PA-824 + 1200 mg QD Linezolid | Total
Number analyzed (Participants) | 53 | 56 | 44 | 65 | 109
events
  Nervous System Disorders | 94 | 83 | 75 | 102 | 177
  #Peripheral Neuropathy | 68 | 56 | 51 | 73 | 124
  Headache | 16 | 16 | 15 | 17 | 32
  Dizziness | 3 | 2 | 1 | 4 | 5
  Dysgeusia | 1 | 3 | 1 | 3 | 4
  Chronic Inflammatory Demyelinating Polyradiculoneurpoathy | 0 | 1 | 0 | 1 | 1
  Dizziness Postural | 1 | 0 | 1 | 0 | 1
  Dystonia | 1 | 0 | 0 | 1 | 1
  #Generalized Tonic-Clonic Seizure | 1 | 0 | 1 | 0 | 1
  Migraine | 0 | 1 | 1 | 0 | 1
  #Optic Neuritis | 1 | 0 | 0 | 1 | 1
  #Seizure | 0 | 1 | 1 | 0 | 1
  Sinus Headache | 1 | 0 | 0 | 1 | 1
  Taste Disorder | 1 | 0 | 1 | 0 | 1
  Tension Headache | 0 | 1 | 0 | 1 | 1
  #Syncope | 0 | 2 | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: Day 1 to 24 Months post-End of Treatment.
Description: Adverse events (AEs) collected for all participants who received at least one dose of study treatment. Includes all AEs which started or worsened on or after the first trial drug administration through 14 days after administration.
  All-cause mortality reported for participants through 24 Months post-End of Treatment.
Groups:
- Bedaquiline + PA-824 + 600mg BID Linezolid: bedaquiline 400 mg once daily for 2 weeks then 200mg 3 times per week plus PA-824 200mg once daily plus linezolid 600mg twice daily .
  Bedaquiline: 100mg tablets
  PA-824: 200mg tablets
  Linezolid: Scored 600mg tablets
- Bedaquiline + PA-824 + 1200mg QD Linezolid: bedaquiline 400 mg once daily for 2 weeks then 200mg 3 times per week plus PA-824 200mg once daily plus linezolid 1200mg once daily .
  Bedaquiline: 100mg tablets
  PA-824: 200mg tablets
  Linezolid: Scored 600mg tablets
Arm/Group | Bedaquiline + PA-824 + 600mg BID Linezolid | Bedaquiline + PA-824 + 1200mg QD Linezolid | Total
All-Cause Mortality (participants affected / at risk) | 5/44 | 3/65 | 8/109
Serious Adverse Events (participants affected / at risk) | 13/44 | 6/65 | 19/109
Other Adverse Events (participants affected / at risk) | 44/44 | 65/65 | 109/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bedaquiline + PA-824 + 600mg BID Linezolid (N=44) | Bedaquiline + PA-824 + 1200mg QD Linezolid (N=65) | Total (N=109)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Pulmonary Tuberculosis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Disseminated Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tuberculoma of Central Nervous System (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Lactic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Generalized Tonic-Clonic Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Optic Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Depression Suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Generalized Anxiety Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Optic Neuropaty (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Transaminases Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bedaquiline + PA-824 + 600mg BID Linezolid (N=44) | Bedaquiline + PA-824 + 1200mg QD Linezolid (N=65) | Total (N=109)
Anaemia (Blood and lymphatic system disorders) | 19 (20) | 20 (20) | 39 (40)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 7 (8) | 8 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 6 (6)
Conjunctivitis allergic (Eye disorders) | 3 (3) | 2 (2) | 5 (5)
Visual impairment (Eye disorders) | 0 (0) | 4 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 5 (5) | 11 (11)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 2 (2) | 7 (7)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (6) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 5 (6) | 11 (14)
Dyspepsia (Gastrointestinal disorders) | 6 (7) | 19 (22) | 25 (29)
Gastritis (Gastrointestinal disorders) | 4 (5) | 4 (4) | 8 (9)
Nausea (Gastrointestinal disorders) | 18 (27) | 21 (32) | 39 (59)
Vomiting (Gastrointestinal disorders) | 16 (24) | 21 (35) | 37 (59)
Influenza (Infections and infestations) | 1 (1) | 5 (5) | 6 (6)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 5 (8) | 7 (10)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 15 (23) | 19 (27)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3) | 6 (6)
Alanine aminotransferase increased (Investigations) | 2 (3) | 8 (9) | 10 (12)
Amylase increased (Investigations) | 5 (6) | 4 (4) | 9 (10)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 8 (9) | 9 (10)
Blood urea increased (Investigations) | 4 (5) | 1 (1) | 5 (6)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 6 (6) | 6 (6)
Gamma-glutamyltran sferase increased (Investigations) | 6 (6) | 13 (13) | 19 (19)
Lipase increased (Investigations) | 3 (4) | 2 (2) | 5 (6)
Transaminases increased (Investigations) | 9 (9) | 2 (3) | 11 (12)
Abnormal loss of weight (Metabolism and nutrition disorders) | 2 (2) | 7 (8) | 9 (10)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 15 (20) | 23 (30)
Hyperamylasaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 7 (7)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 8 (8) | 11 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (9) | 13 (15)
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7) | 8 (8)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 5 (5)
Headache (Nervous system disorders) | 15 (15) | 14 (16) | 29 (31)
Neuropathy peripheral (Nervous system disorders) | 9 (14) | 1 (1) | 10 (15)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (30) | 52 (60) | 75 (90)
Insomnia (Psychiatric disorders) | 3 (4) | 3 (3) | 6 (7)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 5 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (8) | 14 (17)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 13 (14) | 17 (18)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 14 (16) | 16 (18)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 16 (18) | 9 (10) | 25 (28)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (4) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 9 (13) | 15 (19)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 7 (9) | 14 (18)
Hypertension (Vascular disorders) | 2 (2) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT02333799/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT02333799/SAP_001.pdf